CLINICAL TRIAL: NCT04009434
Title: Treatment of Concomitant Mitral Regurgitation by Mitral Valve Clipping in Patients With Successful Transcatheter Aortic Valve Implantation
Acronym: MITAVI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technische Universität Dresden (Other)
Collaborators: Zentrum für Klinische Studien Leipzig (Other); University Medical Center Mainz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MITAVI
Record Dates: First submitted 2019-07-03; First posted 2019-07-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Aortic Stenosis; Mitral Regurgitation
Keywords: Aortic Stenosis; Aortic Disease; Transcatheter Aortic Valve Implantation; Mitral Regurgitation; Mitral Valve Regurgitation; Mitral Disease; Mitral valve clipping; MitraClip; Heart Valve Diseases
MeSH Terms: conditions — Aortic Valve Stenosis; Mitral Valve Insufficiency; Aortic Diseases; Disease; Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAVI (Other): Transfemoral transcatheter aortic valve implantation plus optimal standard of care medical therapy
  Interventions: Device: TAVI
- TAVI/MitraClip (Experimental): Transfemoral transcatheter aortic valve implantation, mitral valve clipping plus optimal standard of care medical therapy.
  Interventions: Device: Mitral Valve Clipping; Device: TAVI

INTERVENTIONS:
Device: Mitral Valve Clipping — Patients receive treatment for mitral regurgitation with mitral valve clipping including standard drug therapy.
  Arms: TAVI/MitraClip
Device: TAVI — Transfemoral transcatheter aortic valve implantation plus optimal standard of care therapy.

SUMMARY:
To evaluate whether patients after successful transfemoral transcatheter aortic valve implantation (TAVI), who have concomitant, moderate to severe mitral regurgitation (MR) benefit from an additional treatment of this valve disease as well.

ELIGIBILITY:
Inclusion criteria

* Planned transfemoral TAVI using an Edwards Sapien 3 Transcatheter Heart Valve (or subsequent models)
* Moderate to severe mitral regurgitation
* Symptom status NYHA II-III
* Treatment and compliance with optimal, individually-tailored guideline directed medical therapy for heart failure for at least 30 days before inclusion
* Age ≥ 18 and < 90 years
* Written informed consent

Exclusion criteria

* MR mechanism/anatomy precluding MitraClip therapy
* Groin blood vessels are not eligible for TAVI procedure
* Massive or torrential tricuspid regurgitation
* Patients who cannot tolerate procedural anticoagulation or post procedural anti-platelet regimen.
* Life expectancy < 1 year due to non-cardiac conditions
* LVEF ≤ 25%
* Hypotension (systolic pressure < 90 mmHg) or requirement of inotropic support or mechanical hemodynamic support
* Cardiomyopathy other than dilated cardiomyopathy
* Fixed pulmonary artery systolic pressure > 70 mm Hg
* Any prior mitral valve surgery or transcatheter mitral valve procedure
* Stroke or transient ischemic event within 6 months prior to randomization
* Severe symptomatic carotid stenosis
* Implant or revision of any rhythm management device (CRT or CRT-D) or implantable cardioverter defibrillator within 90 days prior to randomization
* Untreated clinically significant coronary artery disease requiring revascularization
* Any percutaneous cardiac intervention or carotid surgery within the 30 days prior to randomization, or any cardiac surgery within six months prior to randomization.
* Need for any other cardiovascular surgery (other than MV or AV disease)
* Echocardiographic evidence of intracardiac mass, thrombus, or vegetation
* Active endocarditis or active infections requiring current antibiotic treatment
* Any condition making it unlikely that the patient will be able to complete all protocol procedures
* Patient unable to provide written informed consent prior to study enrolment
* Pregnant or nursing women
* Women of child bearing potential
* Current participation in any other interventional clinical trial
* Patients under legal supervision or guardianship Patients placed in an institution by official or court order

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1162 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Death from any cause and heart failure hospitalization | 1 year
  Composite endpoint of time to heart failure hospitalization or death from any cause

SECONDARY OUTCOMES:
Death from any cause | 1, 2, 3, 4 years
  Time from randomization to death from any cause
Need for mitral valve reintervention | 1, 2, 3, 4 years
  Need for mitral valve reintervention
Mitral regurgitation severity | 1 year
  Mitral regurgitation severity at 12 months
6 Minute Walk Test | 1 year
  Change in 6 Minute Walk Test at 12 months
New York Heart Association Functional Class | 1, 3, 6 months and 1, 2, 3, 4 years
  Course of New York Heart Association (NYHA) Functional Class at 1, 3, 6 months and 1, 2, 3, 4 years

OTHER OUTCOMES:
Number of patients with AEs, SAEs. | 1, 2, 3, 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Axel Linke, MD, Principal Investigator — Technische Universitaet Dresden, HEART CENTER
Locations (1):
- Heart-Center Dresden, Dresden, Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided
After publication of the primary objective, the data might be provided to interested scientists on request (e.g. for meta-analyses, health related registers or other scientific questions) in an anonymized way within five years, if the members of the MITAVI-trial group agree.